CLINICAL TRIAL: NCT00351442
Title: Prospective Study of the Determinants of Host Resistance to HIV-1 Infection
Brief Title: Examining Factors That May Influence Resistance to HIV-1 Infection
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Center for HIV/AIDS Vaccine Immunology (Other)
Responsible Party: Sponsor
Other Study IDs: CHAVI 002; 10464 (Registry Identifier: DAIDS-ES)
Record Dates: First submitted 2006-07-11; First posted 2006-07-12 (Estimated); Last update posted 2014-04-09 (Estimated); Status verified 2014-04

CONDITIONS: HIV Infections
Keywords: Host Resistance
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (3):
- 1: Inidividuals who have been exposed to HIV but remain uninfected.
- 2: HIV infected regular sexual partners of Group 1 participants.
- 3: HIV uninfected individuals or couples who have not been exposed to HIV.

SUMMARY:
Some people who are exposed to the HIV-1 virus are capable of either controlling or completely preventing viral infection. Multiple genetic factors may contribute to preventing or controlling HIV-1 infection. The purpose of this study is to analyze the immune system responses of individuals who are exposed to HIV-1 but remain uninfected.

DETAILED DESCRIPTION:
Even with repeated exposure to HIV-1, some individuals appear to be resistant to infection. The exact mechanism of this resistance, however, remains unknown. The relative risk of HIV-1 infection appears to depend on various factors: route of transmission, viral load of the infected donor, nature and extent of exposure, presence of sexually transmitted infections (STIs), and genetic and immunological status of the exposed individual. This last factor may explain the inherent ability of some people to remain uninfected despite repeated exposure to HIV-1.

Immune response in HIV-1 exposed uninfected individuals is sometimes characterized by specific cytotoxic CD8 T cell response without antibody response, suggesting that resistance may, in part, be mediated by HIV-1 specific T cells. Exposed uninfected individuals may also be genetically protected, in which case key genes-possibly linked to immune responses-may lead to resistance to HIV-1. A clearer understanding of the role of an individual's genetic and immune-mediated resistance to HIV-1 infection is needed and will provide important information for advancing preventive HIV vaccine design. The purpose of this study is to examine the immune responses of individuals who have been exposed to HIV-1, but who remain uninfected. Through the use of highly sensitive technology, low level immune responses and viral levels will be evaluated. The study will also compare genetic profiles, exposure characteristics, donor viral load, STIs, and sexual behaviors among all participants. In the infected member of a serodiscordant couple, the HIV-1 virus will be examined and sequenced.

This observational study will last approximately 24 months. Screening will involve at least one visit and will occur at least 8 weeks prior to study entry. Eligible participants will fall into one of three groups:

* Group 1 will include individuals who have been exposed to HIV-1 but who remain uninfected.
* Group 2 will include HIV infected regular sexual partners of Group 1 members.
* Group 3 will include HIV uninfected individuals or couples who have not been exposed to HIV-1.

Study visits will occur every 3 months for a total of 8 visits. At all visits, participants will verify address location, complete standardized questionnaires about sexual behaviors, and receive HIV safe sex counseling and free condoms. Blood and urine will be collected to test for HIV, STIs, and pregnancy. All participants will undergo a review of their medical history and a physical examination, including a genital exam for both males and females and a pelvic exam for females. At selected visits, participants may opt to provide additional samples of urine, saliva, genital secretions, breastmilk, and feces for research purposes. Groups 1 and 3 will have HIV testing at all but the first study visit; Group 2 will have no HIV testing, but will be assessed for CD4 cell count at all study visits. Participants requiring clinical care for the management of HIV or STIs will be either treated at the study site or referred for appropriate care.

ELIGIBILITY:
Inclusion Criteria for Groups 1, 2, and 3:

* Willing to provide adequate location information
* Planning to remain in the area for the duration of the study

Inclusion Criteria for Group 1:

* HIV-1 antibody positive AND nucleic acid test (NAT) or p24 antigen negative
* Report unprotected receptive or insertive vaginal, oral, or anal intercourse with Group 2 partner on at least 12 occasions (St. Mary's cohort) or 25 occasions (MRC/UVRI Uganda cohort) during the 12 months prior to screening; the first sexual exposure with Group 2 partner must have occurred at least 10 months prior to screening

Inclusion Criteria for Group 2 (St. Mary's cohort):

* HIV-1 infected at screening, as determined by enzyme immunoassay and western blot
* Documentation of HIV-1 infection for at least 12 months prior to screening, as determined by enzyme immunoassay and western blot
* Willing to provide clinical information about HIV-1 RNA and CD4 cell count
* Report unprotected receptive or insertive vaginal, oral, or anal intercourse with Group 1 partner on at least 12 occasions during the 12 months prior to screening; the first sexual exposure with Group 1 partner must have occurred at least 10 months prior to screening

Inclusion Criteria for Group 2 (MRC/UVRI Uganda cohort):

* HIV-1 infected, as determined by enzyme immunoassay and western blot
* Report unprotected receptive or insertive vaginal, oral, or anal intercourse with Group 1 partner on at least 25 occasions during the 12 months prior to screening; the first sexual exposure with Group 1 partner must have occurred at least 10 months prior to screening
* HIV-1 infected for at least 12 months prior to screening, as determined by one of the following criteria:

  1. Report a past medical history indicating Herpes zoster infection within the prior 5 years or report a medical history indicating WHO Clinical Staging Criteria for HIV/AIDS of III or IV within the prior 5 years, OR
  2. CD4 cell count no greater than 450/mm3 for females or no greater than 400/mm3 for males
* Report no prior HIV testing, test HIV-1 seropositive at screening, and meet one of the following criteria:

  1. Report a past medical history indicating Herpes zoster infection within the prior 5 years or report a past medical history indicating WHO Clinical Staging Criteria for HIV/AIDS of III or IV in the prior 5 years, OR
  2. CD4 cell count no greater than 450/mm3 for females or no greater than 400/mm3 for males

Inclusion Criteria for Group 3:

* HIV-1 antibody negative AND nucleic acid test (NAT) or p24 antigen negative
* Test negative for Neisseria gonorrhoeae, syphilis, Chlamydia trachomatis, and trichomoniasis (MRC/UVRI Uganda cohort only)
* Report a monogamous relationship of at least 12 months duration prior to screening

Exclusion Criteria for Groups 1, 2, and 3:

* Injection drug use in the 5 years prior to screening
* Any condition that, in the opinion of the investigator, would be unsafe or interfere with the study
* Any obligations that may require long absences from the area

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community sample, including HIV infected individuals and their uninfected partners.
Sampling Method: Non-Probability Sample
Enrollment: 522 (Estimated)
Dates: Start 2007-02; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew J. McMichael, MD, PhD, Study Chair — University of Oxford, Weatherall Institute of Molecular Medicine
Locations (3):
- Uganda Virus Research Institute, MRC/UVRI Uganda Research Unit on AIDS CHAVI CRS, Entebbe, Uganda
- United Kingdom (2):
  - King's College Hosp., Caldecot Ctr. CHAVI CRS, London
  - St. Mary's Hosp. of London, Imperial College School of Medicine, Clinical Trials Ctr. CHAVI CRS, London

REFERENCES:
- [Background] An P, Bleiber G, Duggal P, Nelson G, May M, Mangeat B, Alobwede I, Trono D, Vlahov D, Donfield S, Goedert JJ, Phair J, Buchbinder S, O'Brien SJ, Telenti A, Winkler CA. APOBEC3G genetic variants and their influence on the progression to AIDS. J Virol. 2004 Oct;78(20):11070-6. doi: 10.1128/JVI.78.20.11070-11076.2004. PMID 15452227
- [Background] Kebba A, Kaleebu P, Rowland S, Ingram R, Whitworth J, Imami N, Gotch F. Distinct patterns of peripheral HIV-1-specific interferon- gamma responses in exposed HIV-1-seronegative individuals. J Infect Dis. 2004 May 1;189(9):1705-13. doi: 10.1086/383227. Epub 2004 Apr 19. PMID 15116309
- [Background] Kebba A, Kaleebu P, Serwanga J, Rowland S, Yirrell D, Downing R, Gilmour J, Imami N, Gotch F, Whitworth J. HIV type 1 antigen-responsive CD4+ T-lymphocytes in exposed yet HIV Type 1 seronegative Ugandans. AIDS Res Hum Retroviruses. 2004 Jan;20(1):67-75. doi: 10.1089/088922204322749512. PMID 15000700
- [Background] Missale G, Papagno L, Penna A, Pilli M, Zerbini A, Vitali P, Pieroni G, Urbani S, Uggeri J, Pinheiro S, Rowland-Jones S, Ferrari C. Parenteral exposure to high HIV viremia leads to virus-specific T cell priming without evidence of infection. Eur J Immunol. 2004 Nov;34(11):3208-15. doi: 10.1002/eji.200424889. PMID 15459901
- [Background] O'Brien SJ, Nelson GW. Human genes that limit AIDS. Nat Genet. 2004 Jun;36(6):565-74. doi: 10.1038/ng1369. PMID 15167933